CLINICAL TRIAL: NCT02676492
Title: A Naturalistic Study Investigating Sleep and Cognitive Learning in Children With and Without Tic Disorders
Status: Completed | Type: Observational
Sponsor: King's College London (Other)
Collaborators: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: HR-15/16-2278
Record Dates: First submitted 2016-02-03; First posted 2016-02-08 (Estimated); Last update posted 2017-08-22 (Actual); Status verified 2016-08

CONDITIONS: Tic Disorders
MeSH Terms: conditions — Tic Disorders | interventions — Efficiency

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Tic Disorder: Boys with a diagnosis of Tourette Syndrome (TS) or chronic tic disorder (CTD) aged 11-14 years
  Interventions: Other: Actigraphy to measure sleep duration and efficiency; Other: 'Sleepsuite' novel cognitive learning tasks
- Control: Boys aged 11-14 years without a diagnosis of TS/CTD (i.e. typically developing)
  Interventions: Other: Actigraphy to measure sleep duration and efficiency; Other: 'Sleepsuite' novel cognitive learning tasks

INTERVENTIONS:
Other: Actigraphy to measure sleep duration and efficiency — Actigraphy watch to be worn on participants' wrist for 14 days and nights
Other: 'Sleepsuite' novel cognitive learning tasks — Novel iPad-administered learning tasks, to be completed one evening and the next morning during actigraphy monitoring period.

SUMMARY:
This study will explore the relationship between sleep, learning, cognition, mood and behaviour in children with Tic Disorders (Tourette Syndrome and Chronic Tic Disorder) compared to typically developing peers.

DETAILED DESCRIPTION:
This project explores the relationship between sleep and learning in childhood with tic disorders, such as Tourette syndrome (TS) and chronic tic disorders (CTD).

TS/CTD are movement disorders characterized by repetitive involuntary movements and/or vocalizations called tics. Sleep related problems are commonly reported for children with TS/CTD and may include problems getting to sleep, waking up frequently during the night, early wakening and tic-related movements in sleep. For typically developing children, sleep disturbances have been linked to problems with mood, behaviour and learning. To date, the relationship between sleep and learning has not been explored for children with TS/CTD.

The aim of this project is to investigate whether there is a relationship between sleep efficiency and learning in boys with and without TS/CTD aged 11-14 years.

Sleep efficiency will be measured using a small actigraphy watch, which will collect information about movements during sleep, night time waking and light exposure. Children will be required to wear the watch for 14 days and nights. Before one night of sleep and again the next morning, children will be asked to complete some tasks on an iPad Air to assess learning. These include 1) 'popping' balloons with faces on them according to specific rules (e.g. boys faces, happy faces), 2) learning novel animal names, 3) navigating a 3D maze. Children will also be administered some standard tests to look at level of intellectual functioning, memory and other thinking skills that may contribute to performance on the computerized tasks. Additionally, children and their parents will be asked to complete questionnaires to assess tics, quality of life, mood and behaviour. The findings of this study will help improve understanding of sleep problems for children with tic disorders to aid the development of specific interventions for this group.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Tourette Syndrome or Chronic Tic Disorder (for clinical group)

Exclusion Criteria:

* Diagnosis of Intellectual Disability (i.e. Full Scale IQ (IntellIigence Quotient) below 70), Autism Spectrum Disorder or Depression
* Currently taking medications to support tic, mood and/or behaviour management

Ages: 11 Years to 14 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Students at mainsteam secondary schools, patients of the Tic and Neurodevelopmental (TANDeM) service at the Evelina Children's Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Relationship between sleep efficiency/duration and cognitive learning | 14 days

SECONDARY OUTCOMES:
Cognitive functioning | Within the 14 days of the study
  A range of cognitive measures will be used to assess general level of intellectual functioning and cognitive skills that are hypothesised to contribute to performance on the SleepSuite learning tasks (including memory, attention, visuo-motor co-ordination and phonological awareness).
Mood and behavioural functioning | Within the 14 days of the study
  A range of self- and parent-report questionnaires will be used to measure participants' mood and behaviour and to see whether these relate to the primary outcome measures of sleep and cognitive learning.

CONTACTS AND LOCATIONS:
Overall Officials: Sally Robinson, Principal Investigator — Guy's and St Thomas' NHS Foundation Trust
Locations (1):
- Evelina Children's Hospital, St Thomas' Hospital, London, United Kingdom